CLINICAL TRIAL: NCT05003830
Title: Application of Multi-probe PET/MR Imaging in the Diagnosis and Evaluation of Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-S1208
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; PET/MR
MeSH Terms: conditions — Alzheimer Disease | interventions — Positron-Emission Tomography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AD group: Patients who meet the core clinical diagnostic criteria for Alzheimer's disease as defined by NIA-AA for mild cognitive decline or probable Alzheimer's disease.
  Interventions: Device: PET/MR
- Healthy control group: Age-matched subjects, who are healthy and have no clinically significant related abnormalities in their physical examinations, laboratory tests, vital signs, or ECG. In addition, no first-degree family history of early-onset AD or other neurodegenerative diseases related to dementia.
  Interventions: Device: PET/MR

INTERVENTIONS:
Device: PET/MR — 18F-FDG, 11C-PIB and 18F-PM-PBB3 injection are radiopharmaceuticals used for positron emission tomography (PET) imaging. 18F-FDG dose is about 3.7-5.4 MBq/kg (0.1 -0.15 mCi/kg), and used in the assessment of brain glucose metabolism. 11C-PIB dose is about 5-10mCi, and used in the assessment of amyloid deposition. 18F-PM-PBB3 dose is about 5-10mCi, and used in the assessment of tau deposition. Use PET/MR equipment for simultaneous PET and MR collection.
  Other Names: Positron Emission Tomography/Magnetic Resonance

SUMMARY:
Alzheimer's disease (AD) is the most common cause of cognitive impairment, and its diagnosis requires a comprehensive analysis of the results of medical history, neuropsychological evaluation, imaging and laboratory tests. Among them, it has been widely recognized that amyloid PET imaging is used in the early diagnosis of AD, tau protein PET imaging is used in the assessment of the progression of AD, and the glucose metabolism PET imaging is used in the assessment of nerve damage. MRI can provide structure, blood perfusion, neural network connection damage and other information through multi-sequence scans. With the help of the PET/MR multi-modal imaging platform and multi-probe imaging technology, it can provide more sensitive and accurate imaging information for early diagnosis and disease assessment of AD, and provide a basis for clinical treatment decision-making.

DETAILED DESCRIPTION:
Cognitive impairment is a common neurodegenerative disease. The incidence of Alzheimer's disease (AD) in people over 65 years old is close to 5%, which brings a heavy burden to society. Relying only on medical history and neuropsychological evaluation, the early diagnosis and differential diagnosis of AD are difficult, and further imaging and laboratory tests are needed. This project will use PET/MRI, the most advanced imaging platform, to design a prospective clinical research program, combined with multi-sequence MRI and multi-probe PET imaging, to evaluate suspected or diagnosed AD patients. Through multi-parameter analysis of the structure MRI, function MRI (3D ASL, BOLD, DTI), metabolism PET (18F-FDG) , Aβ (11C-PIB) and tau (18F-PM-PBB3) PET, combined with clinical information, to evaluate the value of multi-modal imaging for early diagnosis and differential diagnosis of AD, to assist the clinic in the adjustment of early intervention measures and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the core clinical diagnostic criteria for Alzheimer's disease as defined by NIA-AA for mild cognitive decline or probable Alzheimer's disease.
* Subjects are able to understand and sign the informed consent voluntarily, with good compliance.

Exclusion Criteria:

* Have contraindications to PET/MR examination.
* Clinically clear history of stroke.
* Have a history of bipolar disorder or depression.
* Patients with severe heart, liver, and kidney dysfunction.
* Pregnant or lactating women.
* Patients refuse to sign the informed consent.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Central China
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Multi-modal PET/MR imaging mode in Alzheimer's disease | 2 years
  Subjects with suspected or confirmed Alzheimer's disease who have completed multi-modal multi-probe PET/MR imaging, compare with healthy control group to determine the image mode of AD.
Correlation between the results of 18F-PM-PBB3 PET/MR imaging and Alzheimer's disease progression. | 2 years
  Analyze the difference in 18F-PM-PBB3 deposition area and quantitative results in patients with different severity of Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, MD,PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu X, Ruan W, Liu F, Liu Q, Gai Y, Su Y, Liang Z, Sun X, Lan X. Characterizing Early-Onset Alzheimer Disease Using Multiprobe PET/MRI: An AT(N) Framework-Based Study. Clin Nucl Med. 2023 Jun 1;48(6):474-482. doi: 10.1097/RLU.0000000000004663. Epub 2023 Apr 24. PMID 37075301